CLINICAL TRIAL: NCT04036669
Title: Foot Bone Mineral Density and Inflammation in Rheumatoid Arthritis
Brief Title: Adipokines as Predictors of Foot Function, Pain, and Disability in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, clinical Professor, King Saud University
Other Study IDs: file ID: RRC-2014-022
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis; Healthy Control
Keywords: rheumatoid arthritis, adipokines, foot function index, f-BMD
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples from all participants were obtained following an overnight fast; serum was separated and stored at -80oC until reused for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients: RA patients ( N=80; BMI= 26.4± 3.96 ) Eighty patients diagnosed with Rheumatoid arthritis according to American Rheumatology Association criteria and radiographic analysis for at least 10 years previously were randomly involved in this study
- Healthy control: A healthy control group ( N=80; BMI=22.3± 1.85) eighty age and sex-matched healthy controls were included in the study following the assignment of informed consent.

SUMMARY:
Significant increase in the levels of serum adiponectin, ADA, and hsCRP was reported in all RA patients compared to controls.

Compared to patients with early RA, the increase in these markers significantly correlated with disease activity (DAS-ESR), lower f-BMD, radiographic scoring, pain, FFI, and functional limitations in patients with established RA.

Adiponectin showed a negative correlation with serum levels of both ADA and hsCRP. By using ROC curve analysis, optimal cut-off values of adiponectin (28.8 µg/ml), ADA (27.3 IU/L), and hsCRP (1.6 mg/L) could be used to estimate early RA in 45 % of the patients. Similarly, using cut-off values of adiponectin (32.8 µg/ml), ADA (26.1 IU/L ml), and hsCRP (2.5 mg/L), established RA could be predicted in 55 % of patients with 98-99% accuracy.

DETAILED DESCRIPTION:
The present study attempts to evaluate the efficacy of adiponectin, ADA, and foot bone mineral density (fBMD) as predictors of the disease progression in patients with rheumatoid arthritis. A total of 80 RA patients and eighty age and sex-matched healthy controls were included in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients who diagnosed with Rheumatoid arthritis according to American Rheumatology Association criteria and radiographic analysis for at least 10 years previously were randomly involved in this study
* Not receiving any drugs affecting the data obtained
* had Normal daily diets

Exclusion Criteria:

* Subjects with obvious ischemic heart disease (angina, myocardial infarction, and lead electrocardiogram abnormalities),
* HCV, HBV, chronic liver and kidney diseases, hypothyroidism.
* Drugs (diuretics; oral contraceptives).

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eighty patients diagnosed with Rheumatoid arthritis according to American Rheumatology Association criteria and radiographic analysis for at least 10 years previously were randomly involved in this study, and eighty age and sex matched healthy controls were included in the study following assignment of informed consent.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Estimation of Foot bone mineral density (f-BMD) | 3 months
  Foot BMD for all RH patients was performed by Dual Energy X-ray Absorptiometry (DEXA) scan method by using a Lunar DPX densitometer originally used to measure bone mass of small animals and modified to suits the measurements of hand BMD. Foot measurements were applied according to previously reported method
Foot Function Index | 3 months
  Foot Function Index (FFI) is pre-validated questionnaire designed efficiently to measure the effects of foot pathologies such as Rheumatoid Arthritis (RA) on foot function in terms of pain, disability and activity restriction. The FFI has three subscales of measurements; pain, disability, and activity limitation with a total of 23 questions and total score of 10. For each patients, record the respective measurements of the FFI three subscales according to the score range (0-10), whereas; patients with no pain (0); mild pain (1-3); moderate pain(4-6), and severe or worse pain (7-10).

SECONDARY OUTCOMES:
Assessment of serum Adiponectin concentration | 3 months
  The concentrations of serum adiponectin (µg/ml) were measured using human ELISA kit (the Bio-Plex Pro Human Diabetes kit) and measured colorimetrically on the Bio-Plex array reader, according to the manufacturers' instructions.
Assessment of serum Adenosine deaminase (ADA) activity | 3 months
  Serum Adenosine deaminase (ADA) activity was measured by colorimetric kit (Tulip diagnostics (P) Ltd, India)